CLINICAL TRIAL: NCT02598453
Title: An Open-Label, Multi-Center Study to Determine Level of Adherence to Monthly Oral or Every Three Month Intravenous Ibandronate Treatment in Post-Menopausal Women With Osteoporosis or Osteopenia, Who Are GI Intolerant of Daily or Weekly Alendronate or Risendronate
Brief Title: PRIOR Study - A Study of Ibandronate (Boniva) in Postmenopausal Women With Osteoporosis or Osteopenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18058
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (2):
- Ibandronate IV (Experimental): Participants will receive ibandronate 3 mg IV once every 3 months
  Interventions: Drug: Ibandronate
- Ibandronate Oral (Experimental): Participants will receive ibandronate 150 milligrams (mg) tablet once monthly
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — Either 150 mg oral tablet once monthly or 3 mg IV injection once every 3 months
  Other Names: Bonviva/Boniva

SUMMARY:
The purpose of this study is to evaluate treatment adherence to different regimens of ibandronate in postmenopausal women with osteoporosis or osteopenia who are intolerant to daily or weekly alendronate or risedronate therapy due to gastrointestinal (GI) side effects. The anticipated time on study treatment is 12 months, and the target sample size is 517 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Women with postmenopausal osteoporosis or osteopenia
* Discontinuation of daily and /or weekly alendronate or risedronate therapy because of GI intolerance (eg, heartburn, acid reflux, stomach upset)

Exclusion Criteria:

* Inability to stand or sit upright for 60 minutes
* Inability to swallow a tablet whole - Hypersensitivity to any component of Boniva
* Malignant disease diagnosed within previous 10 years (except resected basal cell cancer); contraindications for calcium or vitamin D therapy
* Patients who do not fulfill a minimum 3 months wash-out therapy from any previous bisphosphonate therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2005-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who have greater than or equal to (>=) 75 percent (%) adherence using either monthly oral ibandronate or quarterly intravenous (IV) ibandronate | 12 months

SECONDARY OUTCOMES:
Percentage of participants who have an adherence of >= 75% using ibandronate including both switch and non-switch participants | 12 months
Percentage of participants with GI events based on severity | Up to 10 months
Percentage of participants who experienced a change in frequency and number of GI events | Up to 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (56):
- United States (56):
  - Montgomery, Alabama
  - Lake Havasu City, Arizona
  - Paradise Valley, Arizona
  - Pine Bluff, Arkansas
  - San Diego, California
  - Santa Monica, California
  - Tacoma, California
  - Vista, California
  - Beverly Hills, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Ocala, Florida
  - Palm Harbor, Florida
  - West Palm Beach, Florida
  - Augusta, Georgia
  - Coeur d'Alene, Idaho
  - Champaign, Illinois
  - Evansville, Indiana
  - Natchitoches, Louisiana
  - South Portland, Maine
  - Detroit, Michigan
  - Chaska, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Broken Bow, Nebraska
  - Scottsbluff, Nebraska
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - New York, New York
  - West Haverstraw, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Canfield, Ohio
  - Columbus, Ohio
  - Mayfield, Ohio
  - Oklahoma City, Oklahoma
  - Wyomissing, Pennsylvania
  - Loris, South Carolina
  - Mt. Pleasant, South Carolina
  - Sioux Falls, South Dakota
  - Watertown, South Dakota
  - Bristol, Tennessee
  - Dallas, Texas
  - Denton, Texas
  - San Antonio, Texas
  - Seguin, Texas
  - Temple, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Madison, Wisconsin